CLINICAL TRIAL: NCT02621385
Title: An Open-label, Single-sequence Study to Assess the Effect of Multiple Doses of Tradipitant on Cytochrome P450 3A4 Using Midazolam as a Substrate in Healthy Subjects.
Brief Title: Study to Assess the Effect of Multiple Doses of Tradipitant on CYP3A4 Using Midazolam as a Substrate in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Collaborators: Cross Research S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VP-VLY-686-1102
Record Dates: First submitted 2015-11-17; First posted 2015-12-03 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2015-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tradipitant (Experimental): One dose of midazolam followed by tradipitant dosing for days 3-16. Midazolam is also given on day 16
  Interventions: Drug: tradipitant; Drug: Midazolam

INTERVENTIONS:
Drug: tradipitant — test agent
Drug: Midazolam — substrate for drug-drug interaction assessment

SUMMARY:
This study is designed to evaluate the potential effect of administration of tradipitant on CYP3A4 using midazolam pharmacokinetics as markers.

The study will also further characterize the pharmacokinetics of tradipitant.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and acceptance to provide written informed consent;
2. Subjects must be males or females between 18 and 55 years of age, inclusive;
3. Female subjects of childbearing potential must be non-pregnant and non-lactating and have a negative serum or urine pregnancy test at the Screening visit and at Check-in (Days -1) and agree not to attempt to become pregnant during the course of the study. Female subjects of childbearing potential (including peri-menopausal women who have had a menstrual bleeding within 1 year) must be using appropriate birth control (e.g. intrauterine device [IUD], diaphragm or condom with spermicidal jelly or foam or cervical cap) for a period of 35 days before the first dosing, for the duration of the study, and recommended to use it for one month after the last dose. Women are considered to be not of childbearing potential if they have been surgically sterilized (physician-documented hysterectomy or tubal ligation);

   a. Note: Women are not permitted to use hormonal methods of birth control (e.g. oral contraceptives, hormonal intrauterine device [IUD], patch and steroids) and must use another acceptable method of birth control during the study and recommended to use it for one month after the last dose. Women currently taking oral contraceptives will be required to discontinue their regimen at least two weeks prior to first dosing.
4. Subjects with Body Mass Index (BMI) of ≥18 and ≤33kg/m2 (BMI = weight (kg)/ [height (m)]2);
5. Vital signs (after 3 minutes resting in sitting position) which are within the ranges shown below:

   1. Body temperature between 35.0-37.5 °C;
   2. Systolic blood pressure between 90-150 mmHg;
   3. Diastolic blood pressure between 50-95 mmHg;
   4. Pulse rate between 50-100 beats per minute
6. Willing and able to comply with study requirements;
7. Subjects must be in good health as determined by past medical history, physical examination, electrocardiogram, clinical laboratory tests and urinalysis;

Exclusion Criteria:

1. History of recent (within six months) drug or alcohol abuse as defined in DSM IV, Diagnostic Criteria for Drug and Alcohol Abuse or evidence of such abuse as indicated by the laboratory assays conducted during the Screening visit or at Check-in;
2. Any major surgery within three months of Day 1 or any minor surgery within one month;
3. Donation or loss of 400 mL or more of blood within 3 months prior to the Baseline Visit;
4. History or current evidence of cardiovascular, hepatic, hematopoietic, renal, gastrointestinal or metabolic dysfunction judged by the Investigator to be clinically significant;
5. Any condition requiring the regular use of medication;
6. History of intolerance and/or hypersensitivity to drugs including midazolam, tradipitant, or a medications similar to tradipitant and its accompanying excipients within the past two months prior to Day 1;
7. History (including family history) or current evidence of congenital long QT syndrome or known acquired QT interval prolongation;
8. Subjects who are currently considered at suicide risk, any subject who has ever made a suicide attempt, or those who are currently demonstrating active (within the past 6 months) suicidal ideation as deemed by the Columbia Suicide Severity Rating Scale (C- SSRS);
9. History of liver disease and/or positive for one or more of the following serological results:

   1. a positive hepatitis C antibody test (anti-HCV)
   2. a positive HIV (ELISA and Western-to confirm positive finding) test result c. positive hepatitis B surface antigen (HBsAg)
10. Treatment with any drug known to cause major organ system toxicity (e.g., chloramphenicol or tamoxifen) during the 60 days preceding Day 1;
11. Elevated (> 2 times the upper limit of normal) liver function tests (i.e.

    aspartate aminotransferase (AST [SGOT]), alanine aminotransferase (ALT [SGPT]), and total bilirubin);
12. Inability to be venipunctured and/or tolerate venous access;
13. Subjects who have used tobacco products 3 months prior to dosing. Tobacco users will be defined as any subject who reports cigarette, cigar, tobacco, nicotine gum, nicotine patch or electronic cigarette use;
14. Consumption of >1 drink/day of alcohol for females and >2 drinks/day for males, defined according to the USDA Dietary Guidelines 2010 ;
15. Consumption of >5 cups coffee/tea/day;
16. Participation in the evaluation of any investigational product for 3 months before this study. The 3-month interval is calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study;
17. Use of prescription or OTC medications, including herbal products (e.g., St. John's Wort) within 2 weeks of Day 1;
18. Use of any food or beverage containing alcohol, grapefruit or grapefruit juice, apple or orange juice, vegetables from the mustard green family (e.g. kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard) and charbroiled meat within 1 week before Day 1;
19. Abnormal diets (<1600 or >3500 kcal/day), substantial changes in eating habits in the 4 weeks before this study, or vegetarians;
20. Participation in a previous LY686017 or VLY-686/tradipitant trial;
21. Anyone affiliated with the site or sponsor and/or anyone who may consent under duress;
22. Any other sound medical reason as determined by the clinical Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-11; Primary Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Midazolam Area Under the Curve (AUC) | Pre-dose,0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, and 72 hours
Midazolam time to maximal plasma concentration (Tmax) | Pre-dose,0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, and 72 hours
Midazolam maximal plasma concentration (Cmax) | Pre-dose,0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 18, 24, 36, 48, and 72 hours

SECONDARY OUTCOMES:
α-hydroxymidazolam area under the curve(AUC) | pre-dose, and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours
α-hydroxymidazolam time to maximal plasma concentration (Tmax) | pre-dose, and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24
α-hydroxymidazolam maximal plasma concentration (Cmax) | pre-dose, and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24
Tradipitant and tradipitant metabolites area under the curve (AUC) | pre-dose, and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24
Tradipitant and tradipitant metabolites time to maximal plasma concentration (Tmax) | pre-dose, and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24
Tradipitant and tradipitant metabolites maximal plasma concentration (Cmax) | pre-dose, and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24
Safety of multiple oral doses of tradipitant alone and in combination with midazolam by spontaneous reporting of AEs measured by events related to treatment. | 19 days
Safety of multiple oral doses of tradipitant alone and in combination with midazolam by number of participants with abnormal laboratory values | 19 days
Safety of multiple oral doses of tradipitant alone and in combination with midazolam by number of participants with abnormal ECG values | 19 days
Safety of multiple oral doses of tradipitant alone and in combination with midazolam by number of participants with abnormal vital signs | 19 days
• The Columbia Suicide Severity Rating Scale will be used to assess suicidal behavior and ideation | Baseline, Day 10, Day 19

CONTACTS AND LOCATIONS:
Overall Officials: Milko Radicioni, MD, Principal Investigator — CROSS Research SA
Locations (1):
- Vanda Investigational Site, Arzo, Switzerland